CLINICAL TRIAL: NCT04328766
Title: An Open-Label, Multiple-Dose Clinical Trial to Evaluate the Safety/Tolerability and Pharmacokinetic Interaction Between DWP14012 and DWC202005 in Healthy Volunteers
Brief Title: Pharmacokinetic Interaction Between DWP14012 and DWC202005 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWP14012106
Record Dates: First submitted 2020-03-24; First posted 2020-03-31 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Drug-drug Interaction
MeSH Terms: interventions — Single Person; fexuprazan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DWP14012 Cohort A (Experimental)
  Interventions: Drug: DWC202005, alone
- DWP14012 Cohort B (Experimental)
  Interventions: Drug: DWP14012 + DWC202005
- DWP14012 Cohort C (Experimental)
  Interventions: Drug: DWP14012 + DWC202005, after multiple doses of DWP14012

INTERVENTIONS:
Drug: DWC202005, alone — DWC202005, as a single dose
  Arms: DWP14012 Cohort A
Drug: DWP14012 + DWC202005 — DWP14012 and DWC202005, as a single dose
  Arms: DWP14012 Cohort B
Drug: DWP14012 + DWC202005, after multiple doses of DWP14012 — DWP14012 and DWC202005, after multiple oral doses of DWP14012 once daily for 12 days
  Arms: DWP14012 Cohort C

SUMMARY:
An open-label, multiple-dose clinical trial to evaluate the safety/tolerability and pharmacokinetic interaction between DWP14012 and DWC202005 in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 19 to 50 years with BMI between 18.5 kg/m2 and 30.0 kg/m2
* Capable of understanding provided information and complying with protocol requirements
* Provide written informed consent to participate in the study

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-09-06 (Actual); Primary Completion 2020-11-21 (Actual); Study Completion 2020-11-21 (Actual)

PRIMARY OUTCOMES:
Area under the plasma drug concentration-time curve | upto 48 hours postdose
  AUClast of DWC202005
Peak Plasma Concentration (Cmax) | upto 48 hours postdose
  Cmax of DWC202005
Incidence of Treatment-Emergent Adverse Events | up to 19 days

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network (QPharm), Queensland, Queensland, Australia